CLINICAL TRIAL: NCT06603753
Title: Use of Serum Bilirubin/Albumin Ratio for Early Prediction of Bilirubin Induced Neurological Dysfunction
Brief Title: Role of Serum (B/A) Ratio Compared to (TSB) for Early Prediction of Bilirubin-induced Neurological Dysfunction (BIND).
Status: Not yet recruiting | Type: Observational
Sponsor: alaa aboelhassan mohamed aboelhassan (Other)
Responsible Party: Sponsor-Investigator, alaa aboelhassan mohamed aboelhassan, Assistant Lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: B/A ratio to predict of bind
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hyperbilirubinemia, Neonatal
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to evaluate serum bilirubin/albumin (B/A) ratio compared to total serum bilirubin (TSB) for early prediction of bilirubin-induced neurological dysfunction (BIND).

DETAILED DESCRIPTION:
Introduction Neonatal hyperbilirubinemia is a common problem in neonates. Approximately 60% of term and 80% of preterm babies develop jaundice in the first week of life and about 10% of breastfed babies are still jaundiced at 1 month.

Jaundice due to either indirect (unconjugated) or direct (conjugated) bilirubin within the first 24 h of life should be taken seriously. Early identification and proper management are needed to prevent the serious neurological complications .

When the total serum bilirubin (TSB) rises above the 95th percentile for age (high-risk zone), entry of unconjugated bilirubin into the brain can cause both short-term and long-term neurological dysfunctions (bilirubin encephalopathy) . The increased level of bilirubin is detrimental for nervous system, especially damage the basal ganglia, cerebellum, and brainstem, thus, resulting in bilirubin-induced neurological dysfunction (BIND) .

Bilirubin-induced neurologic dysfunction (BIND) is the term applied to the spectrum of neurologic abnormalities associated with hyperbilirubinemia. It can be further divided into characteristic signs and symptoms that appear in the early stages (acute) and those that evolve over a prolonged period (chronic) . Signs and symptoms of BIND include tone abnormalities such as hypotonia, hypertonia, retrocollis and opisthotonos, in association with varying degrees of drowsiness, lethargy, decreased feeding and irritability .

BIND was also associated with Kernicterus leading to devastating disability including athetoid cerebral palsy, speech and hearing impairment. BIND in neonates is a significant cause of death or lifelong disability, including cerebral palsy (CP) and auditory disorders .

The earliest signs and symptoms of BIND are nonspecific therefore may be easily missed thus an early diagnostic tool is required. BIND score is a scoring system, in which characteristics of mental state, muscle tone, and cry are grouped into three levels of increasing abnormality: stage IA, minimal signs; stage IB, progressive but reversible with treatment; stage II, advanced and largely irreversible, but may be significantly decreased by treatment .

The pathogenesis of BIND is multifactorial and includes interaction between the level of unconjugated bilirubin, free bilirubin, bilirubin bound to albumin, bilirubin passed through brain blood barrier and nerves damage. Although 99.9% of unconjugated bilirubin in the circulation is bound to albumin, a relatively small fraction (only less than 0.1%) remains unbound (free bilirubin) and it can go into the brain across an intact blood brain barrier (BBB) .

There is currently no method available for measuring free bilirubin concentrations accurately in plasma or serum; therefore, adjunct measurements of albumin concentration and bilirubin albumin ratio (B/A) may provide more insight into the likelihood of bilirubin-induced encephalopathy. The B/A ratio is considered a surrogate parameter for free bilirubin and an interesting additional parameter in the management of hyperbilirubinemia. Few studies suggested the utilization of B/A ratios as a predictor for bilirubin-induced neurotoxicity .

ELIGIBILITY:
Inclusion Criteria:• Neonates with hyperbilirubinemia reached level of phototherapy or exchange transfusion according to the American Academy of Pediatrics guidelines [14].

* Age: from 1 to 28 day.
* Full term and preterm babies.
* Both sexes.

Exclusion Criteria:

* Conjugated hyperbilirubinemia.
* Perinatal asphyxia.
* Patients with encephalopathy due to causes other than hyperbilirubinemia.
* Severe birth defects or congenital anomalies.
* Hemodynamic instability.
* Septic patients.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Assiut university children hospital Prospective descriptive study
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Early detection of cases of severe neonatal jaundice for exchange transfusion to avoid complications of kernicterus | baseline
  * The Bind score will be used. The BIND score includes 3 categories: mental status, muscle tone, and cry patterns. Each category will be given a score ranging from 0 to 3.
  * A BIND score of 7-9 will represent advanced signs of encephalopathy, Score of 4-6 will represent moderate signs of encephalopathy and Score of 1-3 encephalopathy subtle signs.
  Laboratory methods:
  * Blood sampling: venous blood will be obtained from each patient under aseptic conditions and collected into 3.2% sodium citrate tubes, except for CBC samples which will be drawn into EDTA tubes.
  * Complete blood count and reticulocyte count: The CBC and reticulocyte counts for both mothers and their babies will be analyzed using an automated hematology analyzer. The CBC parameters analyzed will include hemoglobin level, RBCs, WBCs, and platelet count.
  * Blood Grouping: Blood groups will be detected for both mother and her baby.
  * Liver function tests: The tests will include serum levels of AST, ALT, total bilirubin,

SECONDARY OUTCOMES:
Avoidance of complications of severe neonatal jaundice | baseline
  * Personal data including age and sex, demographics including residence and socioeconomic status.
  * Clinical data including vital signs, body mass index (BMI) and the BIND score.
  * Laboratory data including Complete blood count and reticulocyte count, blood grouping for mother and baby, liver and bilirubin to albumin ration

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud A Ahmed, Dr, Study Director — Assiut University; Jaafar I Mohamad, Prof, Study Director — Assiut University

REFERENCES:
- [Background] Karimzadeh P, Fallahi M, Kazemian M, Taslimi Taleghani N, Nouripour S, Radfar M. Bilirubin Induced Encephalopathy. Iran J Child Neurol. 2020 Winter;14(1):7-19. PMID 32021624
- [Background] Hameed NN, Hussein MA. BIND score: A system to triage infants readmitted for extreme hyperbilirubinemia. Semin Perinatol. 2021 Feb;45(1):151354. doi: 10.1016/j.semperi.2020.151354. Epub 2020 Dec 1. PMID 33309176
- [Background] Paar M, Fengler VH, Reibnegger G, Schnurr K, Waterstradt K, Schwaminger SP, Stauber RE, Oettl K. Determination of binding characteristics as a measure for effective albumin using different methods. Biochim Biophys Acta Gen Subj. 2023 Sep;1867(9):130427. doi: 10.1016/j.bbagen.2023.130427. Epub 2023 Jul 15. PMID 37454915
- [Background] Wang Y, Sheng G, Shi L, Cheng X. Increased serum total bilirubin-albumin ratio was associated with bilirubin encephalopathy in neonates. Biosci Rep. 2020 Jan 31;40(1):BSR20192152. doi: 10.1042/BSR20192152. PMID 31950971
- [Background] El Houchi SZ, Iskander I, Gamaleldin R, El Shenawy A, Seoud I, Abou-Youssef H, Wennberg RP. Prediction of 3- to 5-Month Outcomes from Signs of Acute Bilirubin Toxicity in Newborn Infants. J Pediatr. 2017 Apr;183:51-55.e1. doi: 10.1016/j.jpeds.2016.12.079. Epub 2017 Jan 25. PMID 28131490
- [Background] Ding Y, Wang S, Guo R, Zhang A, Zhu Y. High levels of unbound bilirubin are associated with acute bilirubin encephalopathy in post-exchange transfusion neonates. Ital J Pediatr. 2021 Sep 15;47(1):187. doi: 10.1186/s13052-021-01143-z. PMID 34526082
- [Background] Kang W, Yuan X, Zhang Y, Song J, Xu F, Liu D, Li R, Xu B, Li W, Cheng Y, Zhu C. Early prediction of adverse outcomes in infants with acute bilirubin encephalopathy. Ann Clin Transl Neurol. 2020 Jul;7(7):1141-1147. doi: 10.1002/acn3.51077. Epub 2020 Jun 4. PMID 32495505
- [Background] Kasirer Y, Kaplan M, Hammerman C. Kernicterus on the Spectrum. Neoreviews. 2023 Jun 1;24(6):e329-e342. doi: 10.1542/neo.24-6-e329. PMID 37258501